CLINICAL TRIAL: NCT03544190
Title: Psychometric Evaluation of the Chinese Version of the Resilience Scale-10 for Cancer Children
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW18-012
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2020-11

CONDITIONS: Cancer Childhood
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to translate the original English version of Resilience Scale for Children (RS10) into traditional Chinese. It will then test the psychometric properties of the newly translated RS10.

DETAILED DESCRIPTION:
It has been well documented that cancer and its treatment may have adverse effects on the physical and psychological well-being of children with cancer. Such adverse effects may start from diagnosis and continue for months or even years after the completion of therapy. Cancer and its treatments may also have long-term effects on the psychological well-being of children with cancer, such as decreased self-esteem, increased anxiety and depression that can adversely affect their quality of life.

Numerous studies indicated that resilience effectively prevents the development of mental health problems and is associated with positive mental health outcomes in children and adolescents, such as reduced levels of anxiety, depression and obsessive compulsive symptoms. Assessing resilience in children with cancer is therefore crucial for a thorough understanding of their responses to stress and adversity, which is an essential prerequisite for the design of an appropriate psychological intervention to enhance their resilience and foster the development of their coping mechanisms and positive mental well-being.

This study aims to translate the original English version of Resilience Scale for Children (RS10) into traditional Chinese. It will then test the psychometric properties of the newly translated RS10. In addition, the factorial structure of RS10 will be examined using confirmatory factor analysis (CFA).

ELIGIBILITY:
Inclusion Criteria:

1. ages between 7 and 14;
2. diagnosed with cancer within the previous 6 months and currently undergoing active treatments;
3. able to speak Cantonese and read Chinese.

Exclusion Criteria:

- Those children with cognitive and learning problems identified from their medical records will be excluded.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children should be ages between 7 and 14; diagnosed with cancer within the previous 6 months and currently undergoing active treatments, and able to speak Cantonese and read Chinese.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Resilience level | Baseline
  The Resilience Scale for Children (RS10) was developed to measure a child's capacity to respond to the life changes. The RS10 measures the child's resilience capacity along five core elements: (1) Sense of purpose and meaning, (2) Authenticity, (3) Equanimity, (4) Self-Reliance, and (5) Perseverance.

SECONDARY OUTCOMES:
Number of depressive symptoms | Baseline
  The subjects' depressive symptoms will be assessed using the Chinese version of the CES-DC. The CES-DC comprises 20 fully standardized items to evaluate depressive symptoms. All items are evaluated on a four-point self-report scale in relation to their incidence during the last week, which were scored from 0 to 3, with total possible scores ranging from 0 to 60, with higher scores indicating greater symptomatology.
Levels of self-esteem | Baseline
  The subjects' self-esteem will be assessed using the Chinese version of the RSES. The RSES is designed to measure the global self-esteem of children and adolescents. The scale comprises 10 items, rated using a 4-point Likert scale ranging from 1 to 4, with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Oi Kwan Joyce Chung, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung JOK, Li WHC, Wei X, Cheung AT, Ho LLK, Chan GC. Translation and psychometric evaluation of the Chinese version of the resilience scale for children with cancer. Health Qual Life Outcomes. 2021 Oct 2;19(1):232. doi: 10.1186/s12955-021-01865-y. PMID 34600543